CLINICAL TRIAL: NCT05175534
Title: Contributions of Transesophageal Echocardiography During Episodes of Hemodynamic Instability in Liver Transplant Surgery
Brief Title: Contributions of Transesophageal Echocardiography in Liver Transplant Surgery
Status: Completed | Type: Observational
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PR(AG)511/2019
Record Dates: First submitted 2021-12-08; First posted 2022-01-03 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Liver Transplant; Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: monitoring — peroperative transesophageal echocardiography for monitoring in liver transplant surgery

SUMMARY:
The goal of this study is to describe the safety and impact of transesophageal echocardiography in instability episodes during liver transplantation, especially during reperfusion stage.

After institutional review board approval, this study was performed in Vall d´Hebron University Hospital including patients undergoing liver transplantation Interventions: peroperative transesophageal echocardiography A transesophageal echocardiography scan was performed in case of hemodynamic instability episodes, and immediately after vascular unclamping.

The investigators registered percentatge of patients with diastolic/systolic dysfunction, hypovolemia, vasodilatation, embolism and percentatge of patients with postreperfusion syndrome

DETAILED DESCRIPTION:
A TEE scan was performed in case of hemodynamic instability episodes defined by a decrease of 30% of the mean arterial pressure (MAP) during at least 1 min, and in all patients during immediate graft reperfusion phase and up 30 minutes.

The instability hemodynamic state was classified into four categories: diastolic failure, systolic failure, hypovolemia and vasodilatation.

The diastolic evaluation was performed at ME 4C view using pulsed doppler of the mitral and tricuspid valve at the level of the leaflet tips and tissue Doppler motion of the mitral and tricuspid annulus. The systolic evaluation was performed using tissue Doppler motion of the mitral and tricuspid annulus evaluating S´. Hypovolemia was registered such low filling pressures (mitral lateral E/e´<10 m/s), cardiac index < 2.5 l . min-1 . m-2 and close approximation of the papillary muscles in the TG Mid SAX view. Vasodilatation was registered such low filling pressures (mitral E/e´< 10 m/s) and CI >2.5 l. min-1 . m-2).

An assessment of cardiac filling volumes and contractility, were obtained at two levels: the mid-esophageal four-chamber view (ME 4C) to evaluate the interaction of left and right ventricles and detect possible venous air embolism; and in the trans-gastric mid short axis view (TG mid SAX), to evaluate left ventricular size for the diagnosis of hypovolemia secondary to hemorrhage or altered venous return due to surgical maneuvers on the liver, and segmental wall motion. If the TG mid SAX view was not possible due to the posterior retraction of the stomach during surgery, the ME 4C view, mid-esophageal two chamber view (ME 2C) and mid-esophageal long axis view (ME LAX) was used for the diagnosis of left ventricle systolic dysfunction, and mid-esophageal bicaval view (ME bicaval) was used for the volemia evaluation.

ELIGIBILITY:
Inclusion Criteria: patients undergoing liver transplantation

-

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing liver transplantation
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2016-01-30 (Actual); Primary Completion 2020-05-10 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
determine the cardiac alterations observed during reperfusion phase | during liver transplant
  relationship between cardiac dysfunction and development of post reperfusion syndrome

SECONDARY OUTCOMES:
determine the cardiac alterations during episodes of hemodynamic instability | during liver transplant
  hemodynamic instability was defined as a decrease in the mean arterial pressure (MAP) ≥ 30% from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Susana González-Suárez, MD, PhD, Principal Investigator — Vall d´Hebron University Hospital
Locations (2):
- Spain (2):
  - Susana González Suárez, Barcelona, Catalonia
  - Vall d´Hebron Research Institute VHIR, Barcelona

REFERENCES:
- [Derived] Gonzalez-Suarez S, Corbett M, Hernandez-Martinez A. Impact of graft reperfusion on cardiac function assessed by transesophageal echocardiography during liver transplantation: an observational retrospective study. J Clin Monit Comput. 2024 Apr;38(2):301-311. doi: 10.1007/s10877-023-01110-5. Epub 2023 Nov 30. PMID 38032448